CLINICAL TRIAL: NCT00474513
Title: A PET Study Using [11C] GSK189254 to Establish the Dose, Plasma Concentration and Brain Receptor Occupancy Relationship of GSK239512, a Histamine H3 Antagonist, in Healthy Subjects
Brief Title: An Imaging Study to Investigate the Distribution of GSK239512 in the Brain.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H3B106026
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Mild Cognitive Impairment; Dementia
Keywords: AD, H3, Brain, Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — GSK239512

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK239512

SUMMARY:
GSK239512 is being developed for the treatment of symptoms of cognitive impairment in many diseases. GSK239512 is a drug that binds to the Histamine 3 receptor (a protein) in the brain (receptor occupancy). This study will use the technique of positron emission tomography (PET) as an imaging tool to highlight areas of the brain that GSK239512 has penetrated, and subsequently bound to receptors, after receiving an oral dose of the drug. It will also look at the rate the drug dissociates from the receptors in the brain. Results from the study will provide information on doses of the drug to be given in further studies.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 35 to 49 inclusive at the screening visit.
* Healthy, defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family history), physical examination, laboratory studies, and other tests as judged by the investigator.
* Body weight ≥ 50 kg and BMI within the range of 19-29 kg/m2, inclusive.
* Normal thyroid function tests as judged by the investigator.
* Willingness of subjects to abstain from sexual intercourse with pregnant or lactating women; or willingness to use adequate contraception the time of the first dose of [11C]GSK189254 until completion of the study and for 84 days following the study.
* Capable of giving informed consent and can comply with the study requirements and timetable.
* The subject must be able to read, comprehend and record information.
* A signed and dated written informed consent is obtained from the subject prior to taking part in the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* The subject must have a QTc<450msec (for males) or <480 msec for subjects with bundle branch block

Exclusion Criteria:

* The subject has used or is using regular prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within fourteen days or five half lives (whichever was the longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication would not have interfered with the study procedures or compromised subject safety. Medications considered to be unlikely to interfere with the study are, thyroid replacement therapy, laxatives, occasional use of vitamin supplements, PRN paracetamol and NSAIDs, prophylactic aspirin.
* The subject had a history of drug or alcohol abuse, or had a positive pre-study urine drug / alcohol screen. Abuse of alcohol is defined as an average weekly intake of greater than 21 units or an average daily intake of greater than three units for males. One unit is equivalent to a half-pint (220 mL) of beer or one (25 mL) measure of spirits or one glass (125 mL) of wine.
* History of heavy use (>10 per day) of tobacco or nicotine-containing products within six months of the start of the study.
* Heavy use of caffeine (>6 cups of caffeinated beverage per day).
* The subject had a history or presence of drug or other significant allergy that, in the opinion of the responsible physician, contra-indicated their participation.
* History or presence of neurological or significant psychiatric disease, such as depressive disorder (as defined by HAD depression score >8) or anxiety disorder (as defined by HAD anxiety score >8) See Appendix 7.
* The subject has a history or presence of gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* The subject has donated blood (450 mL) within the last three months before the study.
* The subject has participated in a clinical study with an investigational or a non- investigational drug or device during the previous three months or has participated in more than three studies in the previous year.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with a significant radiation burden that, in combination with the PET scans, may result in the subject receiving more than 10mSv over the previous 3 years.
* History or presence of neurological or psychiatric conditions (e.g., stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, schizophrenia, major depression etc) that may influence the outcome or analysis of the scan results or compromise subject safety.
* Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI questionnaire.
* History of known or suspected seizures, unexplained significant loss of consciousness or history of significant head trauma with loss of consciousness. Subjects who had febrile seizures in childhood may be included if these have ceased by age 5 and they have had no other type of seizure in their medical history and have not been on anti-epileptic medications.
* Allen's test result leading to concern about the patency of both the radial and ulnar arteries in the wrist that is being used for arterial cannulation.
* Needle phobia or fear of arterial blood sampling.
* A positive HIV-1/2, hepatitis B surface antigen or positive hepatitis C antibody result within 3 months of the start of the study.
* Subjects with a QTc of >500 msec.
* Subjects with a known history or presence of sleep disorders based on investigator review of medical history and symptoms

Ages: 35 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Receptor occupancy in the brain after receiving a dose of GSK239512, measured using calculations from PET images at 4 hours and 24 hours post dose

SECONDARY OUTCOMES:
Safety of drug and concentration of GSK239512 in the blood at various timepoints. Using vital signs and ECG, clinical laboratory assessments and PK sampling.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Toronto, Ontario, Canada